CLINICAL TRIAL: NCT04645316
Title: The Effect of Sevoflurane and Desflurane on Clara Cell Protein on the Lung in Liver Transplant Donors: A Randomized Controlled Clinical Trial
Brief Title: The Effect of Sevoflurane and Desflurane on Clara Cell Protein on the Lung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, nureddin teker, Assistant doctor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: NTeker1
Record Dates: First submitted 2020-11-03; First posted 2020-11-27 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-03

CONDITIONS: Inhalation Anesthesia; Lung Injury
Keywords: Sevoflurane; Desflurane; Clara cells protein
MeSH Terms: conditions — Lung Injury | interventions — Sevoflurane; Desflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sevoflurane (Active Comparator): Sevoflurane will use for anesthesia maintenance for liver donor hepatectomy surgery
  Interventions: Drug: Sevoflurane
- Desflurane (Active Comparator): Desflurane will use for anesthesia maintenance for liver donor hepatectomy surgery
  Interventions: Drug: Desflurane
- Total intravenous anesthesia (Placebo Comparator): Total intravenous anesthesia (propofol/remifentanyl) will use for anesthesia maintenance for liver donor hepatectomy surgery
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — In the sevoflurane group (n = 25), after the induction of anesthesia with 2 mg / kg propofol and 1 µg / kg remifentanyl, rocuronium 0.6 mg / kg will be given for intubation. In this group, the Sevoflurane concentration will be adjusted between 1-2%, the BIS value will be 40-60, and it will be inhaled with an air / O2 mixture to be FiO2: 0.4.
  Arms: Sevoflurane
Drug: Desflurane — In the desflurane group (n = 25), after induction of anesthesia with 2 mg / kg propofol and 1 µg / kg remifentanyl, rocuronium 0.6 mg / kg will be given for intubation. In this group, Desflurane concentration will be adjusted between 6-8%, BIS value will be 40-60 and it will be inhaled with a mixture of air / O2 mixture to be FiO2: 0.4.
  Arms: Desflurane
Drug: Propofol — In the propofol-remifentanyl group (n = 25), rocuronium 0.6 mg / kg will be administered for intubation after 2 mg / kg propofol and 1 µg / kg remifentanil. Maintenance of anesthesia will be adjusted to be between 10 mg / kg / h for the first 10 minutes, 8 mg / kg / h for the following 10 minutes, and then by 6 mg / kg / h propofol infusion, with the BIS value between 40-60. Patients in this group will be inhaled with a mixture of air / O2 to be FiO2: 0.4. Inhalation anesthetics will not be used in this group.
  Other Names: TIVA(propofol-remifentanyl)
  Arms: Total intravenous anesthesia

SUMMARY:
Inhalation anesthesia; It means that the anesthetic drugs taken by the respiratory tract pass into the blood through the lung alveoli, reach the brain tissue, and create an anesthetic effect according to the density in the brain tissue. All inhalation anesthetics affect organ functions to varying degrees. Clara cell has been shown to have cell regeneration, immunomodulatory, anti-inflammatory and antioxidant activity in the bronchial epithelium. It is also thought that some substances accumulated in the respiratory system participate in the detoxification. Clara cell protein acts as a protein marker that indicates the severity of airway injuries after exposure to irritants. In this study, we planned to investigate the effect of inhalation anesthetics on Clara cell protein in liver transplant donors who will undergo hepatectomy surgery.

DETAILED DESCRIPTION:
Inhalation anesthesia is still an important source of chemical hazard in the hospital environment due to its widespread use in operating rooms. Factors affecting the presence of anesthetic gases in the environment; device leakage, ventilation, fresh gas flow, and operation of the air cleaning system. Long-term exposure to anesthetic gases is known to adversely affect the health of employees in the operating room.

Clara cell plays a reliable role as a large bronchiolar progenitor cell that can contribute to cell regeneration in the bronchial epithelium. Thus, it contributes to the protection of the normal epithelium of the distal conductive airways. Additionally, it has been shown to have immunomodulatory, anti-inflammatory, and antioxidant activity. It is thought that some substances accumulated in the respiratory system participate in the detoxification.

Operations of patients undergoing hepatectomy usually take 4-6 hours. Inhalation anesthetics are widely used during this surgery. In this study, we thought to show the effect of long-term inhalation anesthesia exposure by performing this surgery on patients in this group. In this study, we aimed to investigate the effect of sevoflurane and desflurane inhalation anesthetics on clara cell protein in liver transplant donors scheduled for hepatectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* living liver donors

Exclusion Criteria:

* smoking
* under 18 years
* over 65 years
* Patients who refused written informed consent forms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
clara cell protein blood levels | baseline,up to 6 hours
  Hepatectomy surgery usually takes 4-6 hours. The clara cell protein levels (baseline) in the blood of the participants before surgery will be compared with the levels of clara cell protein in the blood that will be taken at the end of the surgery. The change between these levels will be measured by ELISA kit.

SECONDARY OUTCOMES:
mean arterial pressure | Procedure (from beginning of anesthesia induction to extubation at 30-minute intervals)
  Mean arterial pressure will be measured at 30-minute intervals from the start of anesthesia induction to extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Muharrem Ucar, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

REFERENCES:
- [Result] Stripp BR, Reynolds SD, Plopper CG, Boe IM, Lund J. Pulmonary phenotype of CCSP/UG deficient mice: a consequence of CCSP deficiency or altered Clara cell function? Ann N Y Acad Sci. 2000;923:202-9. doi: 10.1111/j.1749-6632.2000.tb05531.x. PMID 11193758